CLINICAL TRIAL: NCT02872181
Title: A Randomized Controlled Trial Evaluating Maternal Tilt During Cesarean Section
Brief Title: An Evaluation of Maternal Position During Cesarean Delivery
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Hartford Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: HartfordH
Record Dates: First submitted 2016-01-25; First posted 2016-08-19 (Estimated); Last update posted 2018-08-01 (Actual); Status verified 2018-07

CONDITIONS: Cesarean Section
Keywords: Maternal Position; Tilt; Left Uterine Displacement; Cesarean Delivery; Cesarean Section
MeSH Terms: interventions — Supine Position

ARMS (3):
- BMI <30 (Experimental): Pregnant women undergoing C/S with BMI <30
  Interventions: Procedure: Supine; Procedure: Left uterine displacement
- BMI 30-40 (Experimental): Pregnant women undergoing C/S with BMI 30-40
  Interventions: Procedure: Supine; Procedure: Left uterine displacement
- BMI >40 (Experimental): Pregnant women undergoing C/S with BMI >40
  Interventions: Procedure: Supine; Procedure: Left uterine displacement

INTERVENTIONS:
Procedure: Supine — Placed in Supine position
Procedure: Left uterine displacement — Placed in 15 degrees left uterine displacement

SUMMARY:
During Cesarean Delivery pregnant women are frequently tilted to the left 15 degress to reduce compression of the major blood vessels by the uterus. Despite this common practice, there is no conclusive evidence to support this practice. In fact it may even be deleterious to have women positioned in this position. The aim of the study is to determine whether or not tilting women to the left during cesarean section (CS) is helpful or detrimental. The authors hypothesize that left uterine displacement of 15 degrees, which is commonly employed, is useless for preventing compression of these blood vessels. To investigate this question, women will be randomly assigned to either be tilted 15 degrees to the left during CS or positioned flat on the table. Fetal acid base status, vasopressor/phenylephrine use, patient satisfaction, maternal complications, and fetal complications will all be collected and compared.

ELIGIBILITY:
Inclusion Criteria:

* term pregnant women with an uncomplicated pregnancy course undergoing scheduled cesarean delivery

  * ≥18 years old
  * ASA 1 and 2 (i.e., patient is completely healthy (1) or has mild systemic disease (2)
  * Able and willing to consent to participate

Exclusion Criteria:

* Males

  * <18 years old
  * maternal cardiac/pulmonary/hematologic disorders/renal failure
  * drug/alcohol/tobacco use during pregnancy
  * essential or pregnancy-induced hypertension
  * diabetes greater than 10 years
  * pre-eclampsia or abruptio placenta
  * <37 weeks gestation
  * hemoglobin < 7 g/dL
  * intrauterine growth retardation
  * fetal distress or fetal anomaly
  * Transverse lie
  * Ruptured membranes
  * Severe polyhydramnios or oligohydramnios
  * Multiple gestation
  * severe scoliosis or kyphosis,
  * uterine abnormalities (e.g., large fibroids, bicornuate uterus)
  * Failed spinal (sensory level < T6 after 15 minutes)
  * need to convert to general anesthesia before delivery

Min Age: 18 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 120 (Estimated)
Dates: Start 2016-04; Primary Completion 2020-05 (Estimated); Study Completion 2020-05 (Estimated)

PRIMARY OUTCOMES:
neonatal base deficit from uterine artery immediately after cesarean delivery of the fetus | One data point will be used. The neonatal gas from the uterine artery immediately after delivery

SECONDARY OUTCOMES:
total phenylephrine use in micrograms prior to delivery | The aggregate of the phenylephrine used immediately after spinal (total of 20 minutes) or until delivery of the baby
APGAR scores of the newborn as assessed by the neonatologist immediately after cesarean delivery | 1 and 5 minute apgar scores of the newborn fetus will be compared

CONTACTS AND LOCATIONS:
Overall Officials: adam sachs, MD, Principal Investigator — Hartford Hospital
Locations (1):
- Hartford Hospital, Hartford, Connecticut, United States